CLINICAL TRIAL: NCT02187224
Title: Progesterone Treatment in Reducing Trauma and Alcohol Induced Craving in Individuals Diagnoses With Alcohol Dependence (AD) and Post-tramatic Stress Disorder (PTSD).
Brief Title: Progesterone Effect on Individuals Diagnoses With AD and PTSD.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1603017361; 24330 (Other: Brain & Behavior Research Foundation)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Dependence; Post-Traumatic Stress Disorder (PTSD)
Keywords: Alcohol Dependence; Post-Traumatic stress disorder (PTSD); Progesterone
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Experimental): For the three days prior to each test day every participant in this arm will receive one progesterone capsule (200 mg. bid) on the first day and 2 progesterone capsules per day for days 2 and 3. On the test day the participant will receive the last progesterone capsule (200 mg.bid). On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant)
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator): For the three days prior to each test day every participant in this arm will receive one placebo capsule on the first day and 2 placebo capsules per day for days 2 and 3. On the test day the participant will receive the last placebo capsule. On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant)
  Interventions: Drug: Placebo (for Progesterone)

INTERVENTIONS:
Drug: Progesterone
  Arms: Progesterone
Drug: Placebo (for Progesterone)
  Arms: Placebo

SUMMARY:
This is a randomized control trial with an anticipated 36 participants diagnosed with post-traumatic stress disorder (PTSD) and comorbid alcohol dependence. Participants will be randomized to receive either progesterone (200 mg. bid) or placebo in identical looking capsules for three days.

One goal of this research study is to test if progesterone is more effective than placebo in reducing craving after exposure to trauma cues and alcohol cues in a laboratory paradigm among men and women with AD and PTSD. We hypothesize that progesterone in comparison to placebo will significantly reduce craving for alcohol in response to trauma cues alone and in combination with alcohol cues in individuals with AD and PTSD.

A second goal is to examine if there are gender differences in progesterone effects on stress and alcohol cue-induced craving. We hypothesize that the effects of progesterone on stress and craving will be stronger in women than in men. Participants will be recruited primarily through advertisement, but also through the clinical facilities at the VA and from other collaborators.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 21 to 60;
2. Current diagnosis of AD and PTSD;
3. Drink regularly are not in an active phase of alcohol withdrawal;
4. Not at risk for suicide;
5. Not taking regularly psychoactive drugs including anxiolytics and antidepressants;
6. For women, have regular menses every 25-35 days.

Exclusion Criteria:

1. Current SCID diagnosis of any psychotic disorder;
2. Substance dependence (other than alcohol and nicotine) in the past 30 days;
3. Current unstable medical condition;
4. Positive test results at more than one baseline appointment on urine drug screens conducted for opiates, cocaine, marijuana, benzodiazepines, and barbiturates; for women, amenorrhea, use of oral contraceptives;
5. Known allergy to progesterone or peanuts (vehicle for micronized progesterone);
6. History of thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or Bleeding disorders, heart disease, diabetes or history of stroke.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healtcase System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Ralevski E, Newcomb J, Pisani E, DeNegre D, Peltier M, Jane JS, Yoon G, Petrakis I. Progesterone Attenuates the Stress Response in Individuals with Alcohol Dependence and Post-Traumatic Stress Disorder - A Pilot Study. J Dual Diagn. 2024 Jan-Mar;20(1):39-51. doi: 10.1080/15504263.2023.2294989. Epub 2024 Feb 1. PMID 38147491

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone All Study Participants: For the three days prior to each test day every participant in this arm will receive one progesterone capsule (200 mg. bid) on the first day and 2 progesterone capsules per day for days 2 and 3. On the test day the participant will receive the last progesterone capsule (200 mg.bid). On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant)
  Progesterone
- Placebo All Study Participants: For the three days prior to each test day every participant in this arm will receive one placebo capsule on the first day and 2 placebo capsules per day for days 2 and 3. On the test day the participant will receive the last placebo capsule . On the test day two scripts will be read one trauma related script (most traumatic experience) and one neutral script (relaxed scene given by participant)
  Placebo (for Progesterone)
Period: Overall Study
Arm/Group | Progesterone All Study Participants | Placebo All Study Participants
Started | 8 | 5
Received Trauma Script First | 1 | 4
Received Neutral Script First | 7 | 1
Completed | 7 | 5
Not Completed | 1 | 0
Not completed — Did not show up for test day | 1 | 0

BASELINE CHARACTERISTICS:
Population: Men and women ages 21 to 60; have current diagnosis of either AUD and comorbid PTSD
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone All Study Participants | Placebo All Study Participants | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (8.1) | 49.4 (11.4) | 48.9 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale of Craving (VASC) Baseline no Script
Description: Visual Analogue Scale of Craving (VASC) is a self-report rating scale using the Likert scale (0 Not at all carving alcohol - 10 Extremely carving alcohol)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Progesterone: For the three days prior to each test day every participant in this arm will receive progesterone.
  Progesterone
- Placebo: For the three days prior to each test day every participant in this arm will receive placebo.
  Placebo (for Progesterone)
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale | 1.29 (0.78) | 0.60 (0.89)

2. Secondary Outcome: State Trait Anxiety Inventory (STAI-6) Baseline no Script
Description: Six-item State-Trait Anxiety Inventory (STAI-6) is a psychological inventory consisting of 6 self-report items on a 4-point Likert scale. The STAI-6 measures state anxiety. Higher scores are positively correlated with higher levels of anxiety. STAI-6 scores are classified as "no or low anxiety" (6-12), "moderate anxiety" (13-18), and "high anxiety" (19-24). (minimum score of 6 to a maximum score of 24)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale | 7.86 (0.911) | 9.60 (1.08)

3. Secondary Outcome: Six-item State-Trait Anxiety Inventory (STAI-6) 10 Minutes (Pre-Script #1)
Description: as for outcome 2
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Progesterone Trauma Script; Progesterone Neutral Script: For the three days prior to each test day every participant in this arm will receive progesterone.
  Progesterone
- Placebo Trauma Script; Placebo Neutral Script: For the three days prior to each test day every participant in this arm will receive placebo.
  Placebo (for Progesterone)
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 6.00 (2.65) | 7.50 (1.32) | 6.50 (0.96) | 5.00 (2.35)

4. Secondary Outcome: Six-item State-Trait Anxiety Inventory (STAI-6) 25 Minutes (Post-Script #1)
Description: as for outcome 2
Time Frame: 25 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 11.00 (2.75) | 16.25 (1.38) | 6.17 (0.60) | 5.00 (1.47)

5. Secondary Outcome: Six-item State-Trait Anxiety Inventory (STAI-6) 40 Minutes (Post-Recovery #1)
Description: as for outcome 2
Time Frame: 40 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 9.00 (0.82) | 14.00 (0.41) | 7.07 (0.87) | 8.00 (2.14)

6. Secondary Outcome: Six-item State-Trait Anxiety Inventory (STAI-6) 65 Minutes (Pre-Script #2)
Description: as for outcome 2
Time Frame: 65 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 6.50 (0.67) | 5.00 (1.64) | 9.00 (3.16) | 9.00 (1.58)

7. Secondary Outcome: Six-item State-Trait Anxiety Inventory (STAI-6) 80 Minutes (Post-Script #2)
Description: as for outcome 2
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 14.17 (2.27) | 18.00 (5.57) | 6.00 (4.36) | 8.50 (2.18)

8. Secondary Outcome: Six-item State-Trait Anxiety Inventory (STAI-6) (STAI-6) 95 Minutes (Post-Recovery #2)
Description: as for outcome 2
Time Frame: 95 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 11.17 (1.96) | 14.00 (4.79) | 8.00 (3.95) | 8.25 (1.97)

9. Primary Outcome: Visual Analogue Scale of Craving (VASC) 10 Minutes (Pre-script #1)
Description: as for outcome 1
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 0.16 (1.73) | 0 (0.97) | 0.81 (0.80) | 0.32 (1.75)

10. Primary Outcome: Visual Analogue Scale of Craving (VASC) 25 Minutes (Post-Script #1)
Description: as for outcome 1
Time Frame: 25 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 2.14 (1.80) | 3.93 (0.97) | 1.14 (0.80) | 0.33 (1.74)

11. Primary Outcome: Visual Analogue Scale of Craving (VASC) 40 Minutes (Post-Recovery #1)
Description: as for outcome 1
Time Frame: 40 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 1.15 (1.75) | 1.92 (0.97) | 1.30 (0.79) | 0.40 (1.60)

12. Primary Outcome: Visual Analogue Scale of Craving (VASC) 65 Minutes (Pre-Script #2)
Description: as for outcome 1
Time Frame: 65 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 0.82 (0.81) | 0.20 (1.90) | 3.19 (1.60) | 0 (0.95)

13. Primary Outcome: Visual Analogue Scale of Craving (VASC) 80 Minutes (Post-Script #2)
Description: as for outcome 1
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 3.15 (0.80) | 2.27 (1.83) | 1.13 (1.81) | 0 (0.98)

14. Primary Outcome: Visual Analogue Scale of Craving (VASC) 95 Minutes (Post-Recovery #2)
Description: as for outcome 1
Time Frame: 95 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 1.81 (0.80) | 4.31 (1.76) | 2.14 (1.79) | 0 (0.97)

15. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) Baseline no Script
Description: Visual Analogue Scale of Anxiety (VASA) is a self-report rating scale using the Likert scale (0 Not at all Anxious - 10 Extremely Anxious)
Time Frame: Baseline
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 7 | 5
units on a scale | 0.64 (0.79) | 3.20 (0.89)

16. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) 10 Minutes (Pre-Script #1)
Description: as for outcome 15
Time Frame: 10 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 0 (1.68) | 1.26 (0.96) | 0.20 (0.80) | 0 (1.78)

17. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) 25 Minutes (Post-Script #1)
Description: as for outcome 15
Time Frame: 25 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 2.82 (1.76) | 7.98 (0.97) | 0.03 (0.80) | 0 (1.79)

18. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) 40 Minutes (Post-Recovery #1)
Description: as for outcome 15
Time Frame: 40 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 0 (1.91) | 4.39 (0.99) | 0.85 (0.81) | 0 (1.95)

19. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) 65 Minutes (Pre-Script #2)
Description: as for outcome 15
Time Frame: 65 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 0.18 (0.81) | 0 (1.94) | 0 (1.90) | 2.15 (0.98)

20. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) 80 Minutes (Post-Script #2)
Description: as for outcome 15
Time Frame: 80 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 3.67 (0.81) | 9.89 (1.99) | 0 (1.90) | 1.90 (0.98)

21. Primary Outcome: Visual Analogue Scale of Anxiety (VASA) 95 Minutes (Post-Recovery #2)
Description: as for outcome 15
Time Frame: 95 minutes
Population: All available data was utilized in the analysis using mixed models
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Progesterone Trauma Script | Placebo Trauma Script | Progesterone Neutral Script | Placebo Neutral Script
Number analyzed (Participants) | 7 | 5 | 7 | 5
units on a scale | 1.68 (0.81) | 9.76 (1.98) | 0 (1.98) | 2.05 (0.99)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Progesterone All Study Participants | Placebo All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT02187224/Prot_SAP_000.pdf